CLINICAL TRIAL: NCT00573950
Title: Effects of Cilostazol on Plasma Adipocytokine and Arterial Stiffness in Type 2 Diabetes Patient With Metabolic Syndrome (Randomized, Double-Blind, Placebo-Controled, Cross-Over Study)
Brief Title: Effects of Cilostazol on Plasma Adipocytokine and Arterial Stiffness
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korea University Anam Hospital (Other)
Responsible Party: Sin Gon, Kim, Korea University Anam Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cilostaar
Record Dates: First submitted 2007-12-13; First posted 2007-12-14 (Estimated); Last update posted 2007-12-14 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus, Type 2; Metabolic Syndrome X
Keywords: cilostazol; Type 2 Diabetes mellitus; Metabolic Syndrome; adipocytokines; arterial stiffness; Pulse wave velocity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — Cilostazol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilostazol (Experimental): cilostazol group
  Interventions: Drug: cilostazol
- Placebo (Placebo Comparator): placebo group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: cilostazol — 50 mg two times a day for 2 weeks and then 100mg two times a day for 6 weeks
  Other Names: pletaal
  Arms: Cilostazol
Drug: Placebo — Placebo tablet comparable to 50mg cilostazol two times a day for 2 weeks and then placebo tablet comparable to 100mg cilostazol two times a day for 6 weeks
  Arms: Placebo

SUMMARY:
Cilostazol is an antiplatelet agent used to reduce the symptoms of intermittent claudication. Cilostazol inhibits phosphodiesterase III (PDE III), which causes it to be a vasodilator and inhibitor of platelet aggregation. Recently there were report of beneficial effect of cilostazol like vasodilation, lipid metabolism, and cytokine production. But there were few clinical studies that support these effects of cilostazol. The purpose of this study is to evaluate the vasodilatory and anti-inflammatory effect of cilostazol presented by PWV and plasma adipocytokines.

ELIGIBILITY:
* Eligible for study: 18 year and above, Gender eligible for study: both Inclusion Criteria:Type 2 diabetes patients with metabolic syndrome criteria of Asian-Pacific ATP III guideline
* Type 2 diabetes (at least 1 criteria below)

  1. fasting blood glucose ≥ 126 mg/dL
  2. postprandial 2hour glucose ≥ 200 mg/dL
  3. random blood glucose ≥ 200 mg/dL with typical diabetes symptoms
* Metabolic syndrome : Asian-Pacific ATP III guideline

  1. Fasting blood glucose ≥ 110 mg/dL, or previously diagnosed type 2 diabetes
  2. systolic and/or diastolic blood pressure ≥130/85 mmHg, or treatment of previously diagnosed hypertension
  3. Triglyceride ≥ 150 mg/dL, or Specific treatment for this lipid abnormality
  4. HDL-cholesterol < 40 mg/dL for men and < 50 mg/dL for women, or Specific treatment for this lipid abnormality
  5. Waist circumference ≥ 90 for men and ≥ 80 for women

Exclusion Criteria:

* Hypertensive patients with the use of ACE inhibitor or ARB
* Hyperlipidemic patients with the use of statin or fenofibrate
* Hepatic dysfunction
* Chronic alcohol or drug abuse
* Renal dysfunction
* Heart failure
* Patients who takes hormone replace therapy or steroid containing drugs
* Patients who take drugs like anticoagulant (warfarin), anti-platelet agent (aspirin, ticlopidin), thrombolytic agent (urikinase, alteplase), prostaglandine E1 , drugs inhibit CYP3A4 or CYP2C19, or drugs become substrate of CYP3A4
* Patients who haves disease influencing the results of the study such as neurologic, digestive and neoplastic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-12; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
The effect on pulse wave velocity (PWV) | 8 weeks

SECONDARY OUTCOMES:
the effect on atherosclerotic and inflammatory markers such as adiponectin, hsCRP | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sin Gon Kim, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea Univerisity Anam Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Kim NH, Kim HY, An H, Seo JA, Kim NH, Choi KM, Baik SH, Choi DS, Kim SG. Effect of cilostazol on arterial stiffness and vascular adhesion molecules in type 2 diabetic patients with metabolic syndrome: a randomised, double-blind, placebo-controlled, crossover trial. Diabetol Metab Syndr. 2013 Jul 26;5(1):41. doi: 10.1186/1758-5996-5-41. PMID 23886346